CLINICAL TRIAL: NCT02841644
Title: Operative and Non-operative Treatment of Traumatic Arthrotomies: A Prospective Observational Study
Brief Title: Operative and Non-operative Treatment of Traumatic Arthrotomies
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 04-15-05E
Record Dates: First submitted 2016-06-27; First posted 2016-07-22 (Estimated); Results first posted 2021-08-03 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-01

CONDITIONS: Traumatic Arthrotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traumatic Arthrotomy- Treated Nonoperatively: Patient diagnosed with traumatic arthrotomy treated nonoperatively.
  Interventions: Other: Non-operatively treated traumatic arthrotomy
- Traumatic Arthrotomy- Treated Operatively: Patient diagnosed with traumatic arthrotomy treated operatively.
  Interventions: Procedure: Operatively treated traumatic arthrotomy

INTERVENTIONS:
Procedure: Operatively treated traumatic arthrotomy — operatively treated traumatic arthrotomy.
  Groups: Traumatic Arthrotomy- Treated Operatively
Other: Non-operatively treated traumatic arthrotomy — non-operatively treated traumatic arthrotomy.
  Groups: Traumatic Arthrotomy- Treated Nonoperatively

SUMMARY:
For the last 70 years, orthopaedic dogma has dictated that all injuries that penetrate the joint capsule require formal irrigation and debridement in the operating room to minimize the risk of developing septic complications. The literature supporting this practice is sparse and stems primarily from wartime injuries that may not be generalizable to the smaller, less contaminated arthrotomies seen in the civilian population. Despite the classical teaching of all traumatic arthrotomies requiring irrigation, debridement, and closure in the operating room, numerous surgeons around the country are beginning to treat small traumatic arthrotomies without surgery. The purpose of this study is to evaluate the cost of treatment as well as incidence of adverse events, such as the development of septic arthritis, in patients undergoing operative and non-operative treatment of traumatic arthrotomies.

DETAILED DESCRIPTION:
Background and Rationale Soft tissue wounds around joints are common injuries that are carefully evaluated to identify intra-articular extension. Wound exploration, imaging, and intra-articular saline load injections are commonly utilized to diagnose the presence of a traumatic arthrotomy. The reason for such diligence is that the treatment is dramatically different for a wound that violates the joint compared to one that does not. As opposed to local wound care for simple soft tissue wounds, traumatic arthrotomies are thought to require formal irrigation and debridement in the operating room to minimize the risk of developing septic arthritis.

Septic Joints An injury that penetrates the joint capsule and synovium violates the body's natural barriers that protect the joint from external pathogens. Microorganisms from the environment may enter the joint by direct inoculation or by contiguous spread through the now perforated barrier. By bringing patients to the operating room for formal irrigation and debridement, orthopaedic surgeons are theoretically attempting to minimize the burden of contamination and repair the body's natural barriers to reduce the risk of developing an intra-articular infection. Septic arthritis is an orthopaedic emergency that can result in severe cartilage damage causing long-term joint pain, stiffness, and potentially auto-fusion. If not dealt with in a timely manner, intra-articular infections can result in significant long-term disability, and in extreme cases, can result in overwhelming sepsis and death.

Orthopaedic Dogma Clearly, minimizing the risk of developing septic arthritis is important to every orthopaedic surgeon. Over sixty years ago, observation of a high rate of septic complications in combat injuries that violated the joint. Since then, orthopaedic dogma has dictated that all injuries that violate the joint necessitate formal irrigation and debridement in order to minimize the risk of infectious complications. The literature on the topic is sparse and stems primarily from wartime observations in which the injuries sustained were commonly associated with high levels of contamination, intra-articular fractures, retained foreign bodies, and delayed treatment. The characteristics of these injuries may limit the generalizability of these observations to the civilian population, especially for small, mildly contaminated arthrotomies without associated fracture or retained foreign body.

To date, no studies have prospectively evaluated the benefits of operative irrigation and debridement of traumatic arthrotomies compared to non-operative observation with antibiotics. A single study published showed that patients with open joint injuries treated with operative irrigation and debridement had an infection rate of 2.1%, a value significantly lower than was previously observed in the non-operative cohort of combat injuries. There is little question that large and heavily contaminated arthrotomies benefit from formal irrigation and debridement, but it is unclear if this benefit can extrapolated to smaller, less contaminated injuries. Nevertheless, orthopaedic surgeons continue to debride and irrigate open joints regardless of the burden of contamination or size of arthrotomy.

Small Arthrotomies are Commonly Missed Injuries In an effort to identify and treat as many traumatic arthrotomies as possible, orthopaedic surgeons began looking for additional techniques to aid in their diagnosis. After it's introduction in 1975, saline arthrograms quickly became the gold standard for the diagnosis of small traumatic arthrotomies. This doctrine was called into question when they showed that saline load arthrograms, as they were commonly performed, had a sensitivity of only 43%. Two years later, it was recommended using 155-ml of saline to diagnose 95% of arthrotomies, a volume more than double what was previous used in clinical practice and not easily tolerated by most patients. Most recently, a study showed a false-negative rate of 67% when using 180-mL of saline for their arthrograms, a volume far beyond what would be tolerated in a conscious patient. Despite missing up to half of all small traumatic arthrotomies for the last 40 years, there has not been an outbreak in patients returning with septic arthritis from missed arthrotomies. The absence of such an occurrence raises the question if it is even necessary to formally debride and irrigate small traumatic arthrotomies in the operating room at a great cost to the patient.

Costs of Arthrotomy Despite the relative dearth of evidence supporting the practice of formally irrigating and debriding all open joint injuries, significant healthcare expenditures and additional risks of general anesthesia are undertaken to address this problem. Although the administration of general anesthesia has become extremely safe, it still carries the risk of serious consequences such as heart attack, stroke, and even death. Patients with multiple medical comorbidities are at an even greater risk of a serious perioperative complication.

In addition to the risks of undergoing anesthesia, there are significant costs associated with any operation. A patient diagnosed with an isolated traumatic knee arthrotomy can expect to leave the hospital with a bill of at least $15,000 based on conservative estimates provided by the Department of Research Finance at Carolinas Medical Center. In an era where healthcare costs are spiraling out of control, determining which interventions are efficacious will be paramount in shaping healthcare resource utilization and maintaining long-term sustainability.

Specific Aims:

1. To compare the cost of medical care in patients with traumatic arthrotomies treated with surgical irrigation and debridement versus non-operative treatment with local wound care.
2. To determine the incidence of developing a septic arthritis in patients with a non-operatively treated traumatic arthrotomy.
3. To determine the incidence of developing a septic arthritis in patients with operative treatment of a traumatic arthrotomy.
4. To determine the need for additional surgery (ex: foreign body removal) in patients with a non-operatively treated traumatic arthrotomy.
5. To provide a description of traumatic arthrotomies successfully treated non-operatively.

Study Design Prospective Multi-center Observational Cohort

ELIGIBILITY:
Inclusion Criteria:

* Any patient 18 and older with a traumatic arthrotomy (of any major joint) confirmed by saline load test
* Direct visualization of a capsular rent or intra-articular contents, or air in the joint on CT or radiographs.

  a. Major Joints Include: i. Knee ii. Elbow iii. Wrist iv. Shoulder v. Hip vi. Ankle

Exclusion Criteria:

* Patients who will have severe problems with maintaining follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient 18 years and older with a traumatic arthrotomy
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - University of Kentucky, Lexington, Kentucky
  - Carolinas Medical Center- Main, Charlotte, North Carolina
  - Greenville Health System, Greenville, South Carolina
  - The University of Tennessee Health Science Center, Memphis, Texas

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] HAMPTON OP Jr. The management of penetrating wounds and suppurative arthritis of the knee joint in the Mediterranean Theater of Operations. J Bone Joint Surg Am. 1946 Oct;28(4):659-80. No abstract available. PMID 21003176
- [Background] Levy AS, Lefkoe TP, Whitelaw GP, Kohler S. Management of penetrating pneumatic nailgun injuries of the knee. J Orthop Trauma. 1991;5(1):66-70. doi: 10.1097/00005131-199103000-00012. PMID 2023046
- [Background] Patzakis MJ, Dorr LD, Ivler D, Moore TM, Harvey JP Jr. The early management of open joint injuries. A prospective study of one hundred and forty patients. J Bone Joint Surg Am. 1975 Dec;57(8):1065-70. PMID 1201988
- [Background] Marvel JE, Marsh HO. Management of penetrating injuries of the knee. Clin Orthop Relat Res. 1977 Jan-Feb;(122):268-72. PMID 837616
- [Background] Lanier WL. A three-decade perspective on anesthesia safety. Am Surg. 2006 Nov;72(11):985-9; discussion 1021-30, 1133-48. doi: 10.1177/000313480607201101. PMID 17120937
- [Background] Botney R. Improving patient safety in anesthesia: a success story? Int J Radiat Oncol Biol Phys. 2008;71(1 Suppl):S182-6. doi: 10.1016/j.ijrobp.2007.05.095. PMID 18406924
- [Background] Wolters U, Wolf T, Stutzer H, Schroder T. ASA classification and perioperative variables as predictors of postoperative outcome. Br J Anaesth. 1996 Aug;77(2):217-22. doi: 10.1093/bja/77.2.217. PMID 8881629
- [Background] Chander S, Coakley G. What's New in the Management of Bacterial Septic Arthritis? Curr Infect Dis Rep. 2011 Oct;13(5):478-84. doi: 10.1007/s11908-011-0201-0. PMID 21785928
- [Background] Tornetta P 3rd, Boes MT, Schepsis AA, Foster TE, Bhandari M, Garcia E. How effective is a saline arthrogram for wounds around the knee? Clin Orthop Relat Res. 2008 Feb;466(2):432-5. doi: 10.1007/s11999-007-0006-5. Epub 2008 Jan 10. PMID 18196428
- [Background] Nord RM, Quach T, Walsh M, Pereira D, Tejwani NC. Detection of traumatic arthrotomy of the knee using the saline solution load test. J Bone Joint Surg Am. 2009 Jan;91(1):66-70. doi: 10.2106/JBJS.G.01682. PMID 19122080
- [Background] Metzger P, Carney J, Kuhn K, Booher K, Mazurek M. Sensitivity of the saline load test with and without methylene blue dye in the diagnosis of artificial traumatic knee arthrotomies. J Orthop Trauma. 2012 Jun;26(6):347-9. doi: 10.1097/BOT.0b013e3182255167. PMID 22215059
- [Derived] McKnight RR, Ruffolo M, Wally MK, Seymour RB, Jeray K, E Matuszewski P, Weinlein J, Hsu JR; Southeast Fracture Consortium. Traumatic Arthrotomies: Do They All Need the Operating Room? J Orthop Trauma. 2021 Nov 1;35(11):612-618. doi: 10.1097/BOT.0000000000002093. PMID 34387570

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively
Started | 60 | 120
Completed | 60 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively | Total
Number analyzed (Participants) | 60 | 120 | 180
Age, Continuous [Median (Full Range); unit: years] | 31 [18 to 75] | 28.6 [17 to 84] | 30.5 [17 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 34 | 51
  Male | 43 | 86 | 129
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cost of Treatments
Description: To compare the cost of medical care in patients with traumatic arthrotomies treated with surgical irrigation and debridement versus non-operative treatment with local wound care. To estimate cost associated with TAs, total charge data was acquired for all patients treated at the lead site.
Time Frame: 12 months
Population: We were unable to obtain total charges from half of our our patient population.
Measure: Median (Full Range); unit: USD
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively
Number analyzed (Participants) | 23 | 67
USD | 1089 [55 to 62,378] | 11,973 [863 to 79,920]

2. Primary Outcome: Complications
Description: Complications were defined as septic arthritis, return to the OR, rehospitalization, and osteomyelitis of the injured joint.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively
Number analyzed (Participants) | 60 | 120
Participants | 4 | 18

3. Secondary Outcome: Comparing 3-Month Change in Veterans RAND 12-Item Health Survey (VR-12) by Treatment Method
Description: The veteran rand 12-tem health survey is used to determine change in health related quality of life to estimate disease burden. It is summarized into two scores, a physical component scores (PCS) (range 0-100) and mental component scores (range- 0-100). Higher score indicate better outcomes.
Time Frame: baseline, 3 months
Population: Missing VR-12 from 69 patients.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively
Number analyzed (Participants) | 28 | 83
score on a scale
  VR-12 Physical Health: Baseline | 49 (6.9) | 48.1 (10.6)
  VR-12 Mental Health: Baseline | 50.7 (11.2) | 51.8 (10.9)
  VR-12 Physical Health: 3 month | 36.9 (11.4) | 32.1 (12.3)
  VR-12 Mental Health: 3 Month | 41.9 (7.4) | 46.8 (8.9)
  VR-12 Physical Health: Difference | -12.2 (12.7) | -16.0 (15.3)
  VR-12 Mental Health: Difference | -8.8 (10.5) | -5.1 (12.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Traumatic Arthrotomy- Treated Nonoperatively | Traumatic Arthrotomy- Treated Operatively
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/120
Other Adverse Events (participants affected / at risk) | 0/60 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02841644/Prot_SAP_000.pdf